CLINICAL TRIAL: NCT05501912
Title: A Phase I, Open-Label, Multicenter, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Cancer Activity of ABM-1310 in Patients With BRAF V600-Mutant Advanced Solid Tumors
Brief Title: A Study of ABM-1310 in Patients With BRAF V600-Mutant Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of the applicant's research and development strategy
Sponsor: ABM Therapeutics Shanghai Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABM1310X1101C
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; BRAF V600 Mutation
Keywords: Melanoma; Non-small Cell Lung Cancer; Cholangiocarcinoma; intracranial solid tumor
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages:
  Dose escalation stage: To determine MTD/RP2D and evaluate the safety and tolerability of ABM-1310 monotherapy.
  Dose expansion stage: To further determine RP2D and evaluate the preliminary efficacy of ABM-1310 monotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy Dose Escalation and Dose Expansion (Experimental): In US studies, dose escalation started at a 25 mg BID dose and subsequent dose-escalation groups included: 50 mg BID, 100 mg BID, 150 mg BID, 225 mg BID and 325 mg BID. In this study, the actual dose escalation will be based on a priming dose one level below the highest safe dose or two levels below the MTD that has been tested in US clinical trials when the enrolment of the China study actually initiates, and subsequent escalated doses may be adjusted as appropriate (e.g., the escalated doses following 150 mg BID in the China study may be adjusted to 200 mg BID, 250 mg BID and 300 mg BID. The actual priming dose and subsequent escalated doses for the China study are determined by the SMC) The dose expansion stage in this study will be initiated at the MTD or the optimal dose determined by the SMC as a fixed dose level (MTD or the optimal dose needs to be reviewed by the SMC and subjects are safe and tolerable at that dose level).
  Interventions: Drug: ABM-1310

INTERVENTIONS:
Drug: ABM-1310 — Dose escalation starting dose will be based on a priming dose one level below the highest safe dose or two levels below the MTD that has been tested in US clinical trials.
  Dose expansion will be initiated at the MTD or the optimal dose determined by the SMC as a fixed dose level.

SUMMARY:
This is a Phase I, Open-Label, Multicenter, Dose Escalation and Expansion Study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of ABM-1310 in patients with BRAF V600-Mutant advanced solid tumors. This study consists of two stages: dose escalation and dose expansion. During the dose escalation stage, a classic "3+3" design will be used to guide dose escalation to determine MTD and RP2D. The dose expansion stage will be initiated at the MTD or the optimal dose determined by the Safety Monitoring Committee (SMC ) as a fixed dose level (MTD or the optimal dose needs to be reviewed by the SMC and subjects are safe and tolerable at that dose level).

DETAILED DESCRIPTION:
This is a Phase I, Open-Label, Multicenter, Dose Escalation and Expansion Study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of ABM-1310 in patients with BRAF V600-Mutant advanced solid tumors. The primary objective of this study is to evaluate the safety and tolerability of ABM-1310 monotherapy, and to determine MTD and RP2D. The study will be conducted in two stages:

Dose escalation stage: The dose escalation will be guided by a "3+3" design. In this study, the actual dose escalation will be based on a priming dose one level below the highest safe dose or two levels below the MTD that has been tested in US clinical trials when the enrolment of the China study actually initiates, and subsequent escalated doses may be adjusted as appropriate (e.g., the escalated doses following 150 mg BID in the China study may be adjusted to 200 mg BID, 250 mg BID and 300 mg BID. The actual priming dose and subsequent escalated doses for the China study are determined by the SMC).

Dose expansion stage: Subjects will begin to receive oral doses of ABM-1310, BID, for 28-day cycles at a fixed dose level (as determined at the dose escalation stage).The dose expansion stage is expected to include the following two cohorts of advanced solid tumors with BRAF V600 mutations:

Cohort 1: primary extracranial solid tumors, subjects with BMs preferentially enrolled, up to 15 patients per tumor type; Cohort 2: primary intracranial solid tumors, N = up to 30 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and voluntarily sign informed consent forms (ICFs).
2. Male and female subjects at the age of ≥18 and ≤80 at the time of screening.
3. Patients with histologically or cytologically-confirmed, locally advanced, or metastatic solid tumors with (a) failure of prior standard therapy, (b) no standard therapy available, or (c) for whom standard therapy is not applicable considered by the patient or treating physician. There is no limit to the number of prior treatment lines. Subjects who were previously treated with BRAF and/or MEK inhibitors are allowed to be enrolled in this study.
4. Documentation of positive BRAF V600 mutation is required for enrollment (the blood BRAF V600 test report is received at the dose-escalation stage). Representative tumor specimens suitable for confirmation of BRAF V600 mutations by retrospective analysis are required (for dose-expansion stage only). It is recommended to provide sufficient fresh/archived tumor tissue samples (formalin-fixed paraffin-embedded tumor specimens [preferred]) or 5-10 available unstained sections of good quality for verification of BRAF V600 mutation status at the central laboratory. For any subject who is unable to provide suitable and adequate tumor specimens, re-biopsy (with controllable safety) can be performed in a non-mandatory manner if it is feasible as assessed by the investigator and the subject gives informed consent; if re-biopsy is impossible or refused by the subject, his/her eligibility for enrollment shall be confirmed by both the investigator and the sponsor.
5. Patients with BMs/primary intracranial solid tumors that are asymptomatic, or that are symptomatic but on a stable or decreasing dose of steroids for at least 2 weeks are eligible for enrollment. The specific criteria are as follows:

   * Subjects with inactive and asymptomatic BMs/primary intracranial solid tumors;
   * Subjects who have active, mild neurological signs and symptoms currently requiring no therapy with steroids, and have no history of epileptic seizure within 2 weeks prior to initiation of treatment;
   * Subjects who have active, neurological signs and symptoms and were on a stable or gradually reducing dose up to 4 mg of dexamethasone (or equivalent) per day within 2 weeks prior to initiation of treatment;
6. Subjects who only have evaluable lesions are allowed to be included for the dose escalation stage. They must have at least one measurable lesion (intracranial or extracranial) as defined by RECIST V1.1 criteria or modified RECIST v1.1 for subjects with BMs or the RANO criteria for subjects with primary intracranial solid tumors during screening at the dose expansion stage. Lesions previously treated with radiotherapy shall not be deemed as target lesions unless significant progression as shown on imaging.

   o For BMs from solid tumors;At least one measurable extracranial lesion is required if the longest diameter of the intracranial lesion is less than 0.5 cm (for dose expansion stage only).Subjects with measurable intracranial lesions of 0.5-3 cm in longest diameter (the lower limit of the longest diameter is defined according to the modified RECIST V1.1 criteria are allowed for the study, and measurable extracranial lesions are not required.Subjects with intracranial lesions > 3 cm in longest diameter are not eligible for the study.
7. ECOG score of 0 or 1 or Karnofsky PS score of ≥ 70.
8. Life expectancy > 3 months.
9. Adequate organ function (no blood transfusion and no use of granulocyte colony-stimulating factor, or other hematopoietic stimulator support within 2 weeks before the first administration of the study drug) confirmed as evidenced by:

   * Absolute Neutrophil Count (ANC) ≥ 1.5×10^9/L;
   * Hemoglobin (Hgb) ≥ 90 g/dl;
   * Platelets (Plt) ≥ 75×10^9/L;
   * AST/ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if liver metastases are present;
   * Bilirubin total ≤ 1.5 x ULN, or bilirubin direct < ULN for patients with bilirubin total levels >1.5 ULN;
   * Serum creatinine < 1.5 x ULN or creatinine clearance > 50 mL/min (as calculated via Cockcroft-Gault formula based on the actual body weight of the subject ;
   * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN for subjects not receiving anticoagulant therapy, and INR is maintained within the standard range of treatment prior to starting study drug for subjects receiving anticoagulant therapy.
10. Hepatitis B virus surface antigen (HBsAg) is negative, or HBsAg is positive but HBV DNA titer is below the lower limit of positive detection of the participating site at screening.

    o HBsAg-positive or HBV-DNA positive subjects shall be managed according to institutional guidelines (anti-HBV therapy, where appropriate, and close monitoring of liver function and HBV-DNA replication shall be performed).
11. Negative hepatitis C virus (HCV) antibody test or positive HCV antibody test at the time of screening followed by a negative HCV-RNA test result.

    o HCV-RNA testing is performed only for subjects with a positive HCV antibody test result.
12. Negative HIV test result at the time of screening.
13. All pre-menopausal women and women with menolipsis < 12 months should have a negative pregnancy test result within 7 days before starting study treatment.
14. Must agree to take sufficient contraceptive methods before initiation of study treatment, during the study, and for at least 3 months after the last dose of the study drug.
15. Subjects who are able to swallow a capsule in whole (without chewing, crushing, or opening).

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Subjects with history of neoplasm malignant within 5 years prior to screening, excluding cured carcinoma in situ of cervix, non-melanoma skin cancer, localized prostate cancer and other tumors/cancers that have undergone radical treatment and shown no signs of disease for at least 3 years (This exclusion criterion is only applicable for dose expansion stage. For the dose escalation stage, any patient with double primary malignant solid tumors who can indeed benefit from this study as confirmed by the investigator is eligible for the screening; however, those with any combined primary hematological malignant tumor shall be excluded).
3. Subjects with intracranial hypertension or associated risks (e.g., intracranial infection, intracranial hemorrhage).
4. Subjects with clinically uncontrolled pleural effusion, pericardial effusion, or ascites who, in the judgement of the investigator, are not eligible for enrollment.
5. Subjects with cancerous meningitis (leptomeningeal disease [LMD]).
6. Subjects with history of symptomatic stroke within 6 months prior to initiation of study treatment.
7. Subjects with epileptic seizure within 14 days prior to initiation of study treatment.
8. Impaired cardiac function or clinically significant cardiovascular disorder, including but not limited to any of the following:

   * Left Ventricular Ejection Fraction (LVEF) < 50% as determined via cardiac ultrasound.
   * Long QT syndrome congenital.
   * QTcF (as corrected via Fridericia formula) ≥ 450 ms (males) or 470 ms (females) at screening.
   * Second-degree type II AV block or third-degree AV block.
   * Unstable angina pectoris within 6 months prior to starting study drug.
   * Acute myocardial infarction within 6 months prior to starting study drug.
   * New York Heart Association (NYHA) Class II or higher heart failure within 6 months prior to study treatment.
   * Ventricular arrhythmias > Grade 2 within 6 months prior to study treatment.
   * Poorly controlled hypertension as defined as systolic blood pressure of >160 mmHg or diastolic blood pressure of > 100 mmHg despite use of antihypertensive medications.
   * Combined with any pulmonary embolism, or presence of any serious deep vein thrombosis on lower extremities that require medical interventions such as vena cava filter insertion at the screening .
9. Poorly controlled diabetes (fasting glucose > 10 mmol/L or Glycosylated Haemoglobin (HbA1c) > 8%) despite standard drug therapy.
10. Subjects with:

    * CTCAE grade 2 or higher unresolved diarrhea, or
    * Impaired gastrointestinal (GI) function or GI diseases that may significantly alter the absorption of ABM-1310 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
11. Previous or current, Grade 2 or higher eye disorder, such as retinal vein occlusion (RVO).
12. Severe chronic or active infections requiring intravenous anti-infective therapy within 2 weeks prior to study treatment, including but not limited infectious complications leading to hospitalization, bacteremia, severe pneumonia, or active tuberculosis.

    o Subjects with local fungal infections of skin or nails are allowed for enrollment. Subjects receiving prophylactic antibiotics (e.g., to prevent urinary tract infections or exacerbations of chronic obstructive pulmonary disease) are eligible for study (except for antibiotics prohibited by the protocol).
13. Subjects with solid organ or hematopoietic stem cell transplant within the past 5 years.
14. Patients receiving chemotherapy, targeted therapy, or immunotherapy within 4 weeks prior to study treatment, including the followings:

    * Receiving nitrosourea or mitomycin-C within 6 weeks prior to study treatment.
    * Receiving fluorouracil or small molecule targeted drug therapy within 5 half-lives or 2 weeks (whichever is longer) prior to study treatment.
    * Receiving Chinese herbal or patent medicine within 2 weeks prior to study treatment for anti-tumor indications.
15. Subjects receiving radical radiotherapy or radiotherapy to more than 30% of bone marrow or whole-brain radiotherapy (WBRT) within 4 weeks or palliative radiotherapy for non-target lesions with the aim of relieving symptoms (e.g., bone radiotherapy for pain relief) or stereotactic radiosurgery (including SRS) within 2 weeks prior to starting study drug.
16. Adverse reactions resulted from prior antitumor therapy that have not resolved to baseline or ≤ grade 1 (CTCAE 5.0), except alopecia or ≤ grade 2 peripheral neuropathy, hypothyroidism stabilized by hormone replacement therapy, etc.
17. Subjects who have undergone major surgery within 4 weeks prior to study treatment or who have not recovered from side effects of such therapy or who are expected to undergo major surgery during study treatment. However, a minimum of 2 weeks recovery time from major surgery to starting study drug is required if in investigator's opinion the patient has recovered from such major surgery.
18. Subjects currently receiving therapeutic doses of warfarin sodium or any other coumarin-derivative anticoagulants.
19. Subjects who have received systemic corticosteroids within 2 weeks prior to starting study drug or who have not recovered from side effects of such treatment, excluding conditions described in inclusion criteria for subjects with BMs.

    Note: subjects with topical, intranasal, or inhaled corticosteroids administered; adrenal replacement steroid doses of ≤ 10 mg/day prednisone or the equivalent given; single-use glucocorticoids administered for prophylaxis of contrast media allergy prior to contrast-enhanced imaging are eligible for the study.
20. Subjects who are currently receiving treatment with medication that has a known risk to prolong the QT interval and cannot either be discontinued or switched to a different medication prior to starting study drug.
21. History of alcohol abuse or addiction within 3 months prior to the first dose.
22. Known, documented or suspected history of drug abuse, expect opioids prescribed for pain relief, etc.
23. Past or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might affect the results of the study, and interfere with the subject's participation and study compliance.
24. Other severe and/or uncontrolled concomitant diseases that could cause unacceptable safety risks or compromise compliance with the study protocol.
25. Other conditions that, in the judgement of the investigator, are inappropriate for enrollment in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | From the enrollment of subjects to the end of Cycle 1 (each cycle is 28 days) or up to treatment discontinuation, whichever occurs first, assessed up to 33 days.
  MTD is defined as the highest dose level at which DLT is observed in ≤ 1/6 subjects at one single dose group
Recommended Phase 2 Dose (RP2D) | From the enrollment of subjects to the end of Cycle 1 (each cycle is 28 days) or up to treatment discontinuation, whichever occurs first, assessed up to 33 days.
  RP2D will be a dose either below or equal to MTD
Dose Limiting Toxicity (DLT) | Single dose PK observation period (5 days) and Cycle 1 (28 days) (33 days in total)
  DLT will be evaluated according to NCI-CTCAE V5.0 criteria
The incidence of treatment-related adverse events AE(s) | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal laboratory values | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal vital signs | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal physical examinations | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal ophthalmic evaluation | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal ECG | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal ECOG | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy
Number of participants with abnormal Karnofsky PS | Up to 28 days from treatment discontinuation
  Safety and tolerability of ABM-1310 monotherapy

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Maximum plasma concentration (Cmax) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Time to maximum plasma concentration (Tmax) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Half-life (T1/2) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Apparent plasma clearance (CL/F) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Apparent volume of distribution (Vz/F) | only 5 days prior to dose escalation stage
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Area under the concentration time curve (AUC) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Maximum plasma concentration (Cmax) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Time to maximum plasma concentration (Tmax) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Half-life (T1/2) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Apparent plasma clearance (CL/F) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Apparent volume of distribution (Vz/F) | Up to Day 1, Day 8, Day 15, Day 22 and Day 28 of Cycle 1. Up to Day 1 and Day 2 of Cycle2. After Cycle2, tests every 2 cycles (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 monotherapy
Objective Response Rate (ORR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Disease Control Rate (DCR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Duration of Response (DOR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Progression free survival (PFS) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Intracranial Objective Response Rate (ORR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary intracranial efficacy of ABM-1310 monotherapy
Intracranial Disease Control Rate (DCR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary intracranial efficacy of ABM-1310 monotherapy
Intracranial Duration of Response (DOR) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary intracranial efficacy of ABM-1310 monotherapy
Intracranial Progression free survival (PFS) | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary intracranial efficacy of ABM-1310 monotherapy
Deepness of Response（DPR） | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary efficacy of ABM-1310 monotherapy
Intracranial Deepness of Response（DPR） | From the enrollment of subjects to the time of disease progression in radiological imaging or death from any cause, whichever occurs first, assessed approximately 12 months.
  Preliminary intracranial efficacy of ABM-1310 monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Shanghai East Hospital
Locations (10):
- China (10):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgeng Hospital, Beijing, Beijing Municipality
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Affiliated Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lake D, Correa SA, Muller J. Negative feedback regulation of the ERK1/2 MAPK pathway. Cell Mol Life Sci. 2016 Dec;73(23):4397-4413. doi: 10.1007/s00018-016-2297-8. Epub 2016 Jun 24. PMID 27342992
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] Wellbrock C, Karasarides M, Marais R. The RAF proteins take centre stage. Nat Rev Mol Cell Biol. 2004 Nov;5(11):875-85. doi: 10.1038/nrm1498. PMID 15520807
- [Background] Lovly CM, Dahlman KB, Fohn LE, Su Z, Dias-Santagata D, Hicks DJ, Hucks D, Berry E, Terry C, Duke M, Su Y, Sobolik-Delmaire T, Richmond A, Kelley MC, Vnencak-Jones CL, Iafrate AJ, Sosman J, Pao W. Routine multiplex mutational profiling of melanomas enables enrollment in genotype-driven therapeutic trials. PLoS One. 2012;7(4):e35309. doi: 10.1371/journal.pone.0035309. Epub 2012 Apr 20. PMID 22536370
- [Background] Fujio S, Juratli TA, Arita K, Hirano H, Nagano Y, Takajo T, Yoshimoto K, Bihun IV, Kaplan AB, Nayyar N, Fink AL, Bertalan MS, Tummala SS, Curry WT Jr, Jones PS, Martinez-Lage M, Cahill DP, Barker FG, Brastianos PK. A Clinical Rule for Preoperative Prediction of BRAF Mutation Status in Craniopharyngiomas. Neurosurgery. 2019 Aug 1;85(2):204-210. doi: 10.1093/neuros/nyy569. PMID 30481321
- [Background] Giunta EF, De Falco V, Napolitano S, Argenziano G, Brancaccio G, Moscarella E, Ciardiello D, Ciardiello F, Troiani T. Optimal treatment strategy for metastatic melanoma patients harboring BRAF-V600 mutations. Ther Adv Med Oncol. 2020 Jun 19;12:1758835920925219. doi: 10.1177/1758835920925219. eCollection 2020. PMID 32612709
- [Background] Schreck KC, Grossman SA, Pratilas CA. BRAF Mutations and the Utility of RAF and MEK Inhibitors in Primary Brain Tumors. Cancers (Basel). 2019 Aug 28;11(9):1262. doi: 10.3390/cancers11091262. PMID 31466300
- [Background] Khalifa J, Amini A, Popat S, Gaspar LE, Faivre-Finn C; International Association for the Study of Lung Cancer Advanced Radiation Technology Committee. Brain Metastases from NSCLC: Radiation Therapy in the Era of Targeted Therapies. J Thorac Oncol. 2016 Oct;11(10):1627-43. doi: 10.1016/j.jtho.2016.06.002. Epub 2016 Jun 23. PMID 27343440
- [Background] Carr S, Smith C, Wernberg J. Epidemiology and Risk Factors of Melanoma. Surg Clin North Am. 2020 Feb;100(1):1-12. doi: 10.1016/j.suc.2019.09.005. Epub 2019 Nov 4. PMID 31753105
- [Background] Chi Z, Li S, Sheng X, Si L, Cui C, Han M, Guo J. Clinical presentation, histology, and prognoses of malignant melanoma in ethnic Chinese: a study of 522 consecutive cases. BMC Cancer. 2011 Feb 25;11:85. doi: 10.1186/1471-2407-11-85. PMID 21349197
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Dienstmann R, Tabernero J. BRAF as a target for cancer therapy. Anticancer Agents Med Chem. 2011 Mar;11(3):285-95. doi: 10.2174/187152011795347469. PMID 21426297
- [Background] Amaral T, Sinnberg T, Meier F, Krepler C, Levesque M, Niessner H, Garbe C. The mitogen-activated protein kinase pathway in melanoma part I - Activation and primary resistance mechanisms to BRAF inhibition. Eur J Cancer. 2017 Mar;73:85-92. doi: 10.1016/j.ejca.2016.12.010. Epub 2017 Feb 3. PMID 28169047
- [Background] Davies MA, Saiag P, Robert C, Grob JJ, Flaherty KT, Arance A, Chiarion-Sileni V, Thomas L, Lesimple T, Mortier L, Moschos SJ, Hogg D, Marquez-Rodas I, Del Vecchio M, Lebbe C, Meyer N, Zhang Y, Huang Y, Mookerjee B, Long GV. Dabrafenib plus trametinib in patients with BRAFV600-mutant melanoma brain metastases (COMBI-MB): a multicentre, multicohort, open-label, phase 2 trial. Lancet Oncol. 2017 Jul;18(7):863-873. doi: 10.1016/S1470-2045(17)30429-1. Epub 2017 Jun 4. PMID 28592387
- [Background] Flaherty KT, Hodi FS, Fisher DE. From genes to drugs: targeted strategies for melanoma. Nat Rev Cancer. 2012 Apr 5;12(5):349-61. doi: 10.1038/nrc3218. PMID 22475929
- [Background] Kaley T, Touat M, Subbiah V, Hollebecque A, Rodon J, Lockhart AC, Keedy V, Bielle F, Hofheinz RD, Joly F, Blay JY, Chau I, Puzanov I, Raje NS, Wolf J, DeAngelis LM, Makrutzki M, Riehl T, Pitcher B, Baselga J, Hyman DM. BRAF Inhibition in BRAFV600-Mutant Gliomas: Results From the VE-BASKET Study. J Clin Oncol. 2018 Dec 10;36(35):3477-3484. doi: 10.1200/JCO.2018.78.9990. Epub 2018 Oct 23. PMID 30351999
- [Background] Sosman JA, Kim KB, Schuchter L, Gonzalez R, Pavlick AC, Weber JS, McArthur GA, Hutson TE, Moschos SJ, Flaherty KT, Hersey P, Kefford R, Lawrence D, Puzanov I, Lewis KD, Amaravadi RK, Chmielowski B, Lawrence HJ, Shyr Y, Ye F, Li J, Nolop KB, Lee RJ, Joe AK, Ribas A. Survival in BRAF V600-mutant advanced melanoma treated with vemurafenib. N Engl J Med. 2012 Feb 23;366(8):707-14. doi: 10.1056/NEJMoa1112302. PMID 22356324
- [Background] Hauschild A, Grob JJ, Demidov LV, Jouary T, Gutzmer R, Millward M, Rutkowski P, Blank CU, Miller WH Jr, Kaempgen E, Martin-Algarra S, Karaszewska B, Mauch C, Chiarion-Sileni V, Martin AM, Swann S, Haney P, Mirakhur B, Guckert ME, Goodman V, Chapman PB. Dabrafenib in BRAF-mutated metastatic melanoma: a multicentre, open-label, phase 3 randomised controlled trial. Lancet. 2012 Jul 28;380(9839):358-65. doi: 10.1016/S0140-6736(12)60868-X. Epub 2012 Jun 25. PMID 22735384
- [Background] Valpione S, Carlino MS, Mangana J, Mooradian MJ, McArthur G, Schadendorf D, Hauschild A, Menzies AM, Arance A, Ascierto PA, Di Giacomo A, de Rosa F, Larkin J, Park JJ, Goldinger SM, Sullivan RJ, Xu W, Livingstone E, Weichenthal M, Rai R, Gaba L, Long GV, Lorigan P. Rechallenge with BRAF-directed treatment in metastatic melanoma: A multi-institutional retrospective study. Eur J Cancer. 2018 Mar;91:116-124. doi: 10.1016/j.ejca.2017.12.007. Epub 2018 Jan 19. PMID 29360604
- [Background] Tietze JK, Forschner A, Loquai C, Mitzel-Rink H, Zimmer L, Meiss F, Rafei-Shamsabadi D, Utikal J, Bergmann M, Meier F, Kreuzberg N, Schlaak M, Weishaupt C, Pfohler C, Ziemer M, Fluck M, Rainer J, Heppt MV, Berking C. The efficacy of re-challenge with BRAF inhibitors after previous progression to BRAF inhibitors in melanoma: A retrospective multicenter study. Oncotarget. 2018 Sep 28;9(76):34336-34346. doi: 10.18632/oncotarget.26149. eCollection 2018 Sep 28. PMID 30344946
- [Background] Becco P, Gallo S, Poletto S, Frascione MPM, Crotto L, Zaccagna A, Paruzzo L, Caravelli D, Carnevale-Schianca F, Aglietta M. Melanoma Brain Metastases in the Era of Target Therapies: An Overview. Cancers (Basel). 2020 Jun 21;12(6):1640. doi: 10.3390/cancers12061640. PMID 32575838
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- See also: CNKI References — http://kns.cnki.net/kcms/detail/detail.aspx?dbcode=CJFD&dbname=CJFDLAST2016&filename=WYSB201608009&uniplatform=NZKPT&v=6C1JD8cdF_QOvutfIkH1DVft0m4rKB6wcvOgXS13Fwm9Pp_DifWR4NKe0xs9dlhT